CLINICAL TRIAL: NCT05133726
Title: Reducing Inpatient Readmission Rates for Patients Discharged From Acute Psychiatric Care in Alberta Using Peer and Text Message Support: Protocol for an Innovative Supportive Program
Brief Title: Peer and Text Message Support to Reduce Readmission Rates for Patients Discharged From Acute Psychiatric Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00111459
Record Dates: First submitted 2021-10-21; First posted 2021-11-24 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Psychiatric Illness
Keywords: Psychiatric Illness; Peer support; Text Message; Electronic health (eHealth); Readmission rate
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Stepped edge design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Text Message cluster (Experimental): This arm will receive only daily text message support for six months plus weekly text message over 6 weeks (six information text messages all together)
  Interventions: Other: Text4Support
- Text message with or without peer support (Experimental): All individuals in this cluster will receive daily text message support for six months plus weekly text message over 6 weeks (six information text messages all together) with some selected members also receiving peer support for six months
  Interventions: Other: Text4Support; Other: Peer support
- Control group (No Intervention): This group will only receive usual care plus weekly text message over 6 weeks (six information text messages all together) with provides information about community services

INTERVENTIONS:
Other: Text4Support — Daily supportive text messages
  Other Names: Supportive messages
  Arms: Text Message cluster; Text message with or without peer support
Other: Peer support — Meeting with peers who have lived experiences with similar diagnoses but are in recovery
  Arms: Text message with or without peer support

SUMMARY:
Avoidable hospital readmissions are a pressing problem for our healthcare system. They lead to substantial human suffering and higher financial costs. Most discharged psychiatric inpatients in Alberta are offered follow-up appointments with Alberta Health Services (AHS) Addiction and Mental Health (AMH) community providers. Patients often wait 28-38 weeks for their first appointment, which leads many to miss their first appointments, and increases the likelihood of relapse. As a result, patients discharged into the community are readmitted to the Emergency Department (ED). To address this significant revolving door, the investigators will implement a low-cost, evidence-based system that delivers daily supportive texts to patients' mobile phones. The text messages developed by experts and service users, based on cognitive behavioral therapy principles. Our proposed program also includes peer support from previous mental health patients who have had similar challenges as participants, but are now in recovery. In this way, the investigators aim to reduce the psychological treatment and support gap for AMH patients who have been discharged from acute care and are scheduled to receive mental health and psychiatric treatment from A&MH services after a long wait. Our pilot test of these interventions provide evidence that psychiatric readmissions, and emergency department visits can be reduced by 10-25% if implemented at scale in Alberta, thus resulting in cost-savings for individuals and the province.

DETAILED DESCRIPTION:
Background & Rational Avoidable hospital readmission is a growing concern in health systems across the world. Readmissions often lead to significant physical, psychological and financial suffering on the part of patients and their families. The health system is also affected by high readmission rates. Infrastructural, human and financial resources, which are limited, often get stretched. This is particularly true in the era of the 2019 corona virus disease (COVID-19) pandemic, which has seen many hospitals overwhelmed by rising emergency presentations. Consequently, there is a renewed interest to seek out solutions to mitigate avoidable readmissions, particularly in acute care.

Patients with psychiatric disorders have the highest early readmission rates among all hospitalized patients. Early readmission is defined as readmission within 30 days of previous discharge. Whereas deinstitutionalization of care and transition to community-based mental health care has been an approach of focus for decades, early hospital readmission remains high. Unmet need for psychological treatment and the limited human resources to address this gap is a major cause of high 30-day readmissions rates in mental acute units.

In Alberta, Canada, about 8.4-11.9% of residents suffer from mental illness, but less than 25% of these patients report that their mental health care needs were fully met. This is despite almost 70% of mental health patients utilizing a provincial mental health service the year before, according to a 2014 mental health gap assessment report. The greatest unmet need cited is the lack of sufficient, accessible, and affordable counselling. Their next greatest concern was an unmet need for tailored information on their own mental health challenges. This is despite the 426 distinct interventions within AHS to address addiction and mental health challenges through community health clinics, and free-standing AMH facilities, among others. Interestingly, 86% of Alberta Health Services direct providers believe that they provide sufficient information to clients. This contradiction between patients and community providers' perspectives reinforces concerns that services may not be well tailored to the diverse perceived needs of various patient groups. A consequence of this gap is the high demand for more specialist services, and high readmissions after discharge from a recent hospital stay with attendant implications on the cost of health services. One study reports 90-day readmission rates of up to 14.0%, with the median time to readmission being 24 days. More findings from the 2014 mental health gap assessment revealed that current management strategies are reactive, with system resources heavily invested in inpatient, residential and crisis services. Technology was noted to be under-utilized in the province. Reducing the felt need for hospital visits by providing alternative effective care will mitigate the existing strain on healthcare human and financial resources due to mental health challenges. To address this challenge, the investigators propose an innovative program which augments peer support from previous mental health patients now in recovery with an evidence-based supportive text messaging developed using the principles of cognitive behavioral therapy (CBT).

Components of the innovation

1. Peer support is valued in recovery-oriented models of mental health and increasingly implemented. Evidence indicates positive effects, including lower inpatient service use, better relationships with providers and increased engagement. Peer Support Workers (PSWs) who are in recovery and have lived experience as former patients will play central roles in this study, including delivering some of the interventions proposed. PSW activities will include supportive face-to-face visits, interactive phone calls/texts/zoom meetings with patients, advocacy, connecting patients with community resources, and experiential sharing. PSWs will be actively engaged through all provincial practice councils, they are embedded within many Alberta addiction and mental health (AMH) programs, making this solution workable. Evidence also shows that peers support may also benefit peer PSWs, enhancing feelings of competence and personal value.
2. Text4Support to be provided through ResilienceNHope online application (https://application.resiliencenhope.com/), is a low cost, evidence-based, supportive text messaging program which will be coupled with or without peer support services to reduce the psychological treatment and support gap for A&MH patients who have been discharged from acute care into community. Starting a day after enrolment, intervention-group patients will receive daily unidirectional (no-reply) supportive text messages. The messages will be written by cognitive behavior therapists in partnership with patients and preprogramed into ResilienceNHope which will deliver the messages to the patients. The Text4Support program was developed based on knowledge from randomized controlled trials conducted in Ireland and Alberta. The program is also based on knowledge from the highly successful award winning Text4Mood program in Alberta's North Zone which improved the psychological treatment gap and was effective, scalable (i.e., > 10,000 recipients within 6 months) and the Text4Hope program launched in Alberta during the COVID 19 pandemic which was also effective and scalable (> 48,000 subscribers within 3 months). Text4Support provides Cognitive Behavioral Therapy (CBT)-based and diagnosis-specific (i.e., mood disorders, anxiety disorders, schizophrenia and other psychotic disorders, substance use disorders, adjustment disorders or personality disorders), daily supportive text messages for 6 months. Some examples of the text messages are:

   * What lies behind you and what lies before you are tiny matters compared to what lies within you. Have faith in yourself, and success can be yours.
   * There are 2 days in the week we should not worry about, yesterday and tomorrow. That leaves today. Live for today.
   * Stumbling blocks can become stepping stones to a better life. You can turn adversities into opportunities. Don't be discouraged by today's problems.
   * Letting go of resentment is a gift you give yourself. It will ease your journey immeasurably. Make peace with everyone, and happiness will be yours.

With respect to content, analysis of Alberta service data suggests that diagnostic clusters for patients discharged from acute into community for follow-up falls into six major categories: mood disorders, anxiety disorders, schizophrenia and other psychotic disorders, substance use disorders, adjustment disorders and personality disorders. Thus, text message content will focus on two dimensions. First, general content that is indicated regardless of symptomatology will be presented, including messages of self-care, social support, hope, affirmation, and recovery. Second, specific content will be provided that focuses on management of symptoms related to the specific conditions described above (e.g., activity scheduling in depression). As a component of scalability and inclusiveness, text message content can also be customized based on end user characteristics. Specifically, the investigators will explore content that is sensitive to needs based on age group, cultural identity, gender identification, and non-English language communication. This serves to enhance access for diverse groups, many of whom may be marginalized or underserved. In addition, patients identified to be most at-risk of readmission to hospital will be offered peer support, which also takes into account age and gender of both the patient and PSWs. Options for matching patients and PSWs by cultural identity and sexual orientation will be explored as the project is scaled up and the pool of PSWs increases. Consequently, recruitment of PSWs will take into account diversity in age, gender, cultural identity and sexual orientation.

Study aim This study is designed to address gaps in care/support available at the community level for psychiatric patients discharged from hospital and referred to community mental health services for follow-up. The investigators aim to reduce the psychological treatment and support gap for AMH patients who have been discharged from acute care and are scheduled to receive mental health and psychiatric treatment from AMH services after a long wait. Our pilot test (unpublished) of these interventions provide evidence that psychiatric readmissions, and emergency department visits can be reduced by 10-25% if implemented at scale in Alberta, thus resulting in cost-savings for individuals and the province.

Methods and analysis This study will both evaluate the effectiveness of this intervention as well as implementation context and outcomes. The Consolidated Framework for Implementation Research (CFIR) will provide an overarching guidance to design, implementation, and evaluation by examining outer/inner contexts, intervention characteristics, and stakeholders involved as well as the process of implementation.

Further, using the Reach-Effectiveness-Adoption-Implementation- Maintenance (RE-AIM) framework, the investigators will: examine the reach of the interventions, i.e., text and peer support; evaluate their effectiveness; gauge support for their adoption; evaluate fidelity in implementation; and document the maintenance (sustainability) of implementation post-trail.

Study design A pragmatic stepped-wedge cluster-randomized approach will be applied, providing Text4Support and Peer Support Service (PSS) to 10,800 patients recruited across 11 acute care sites and day hospitals across Alberta as the clustered unit of randomization. The design reconciles constraints under which policy makers and service managers operate with need for rigorous scientific evaluations. In a stepped-wedge study, the design is extended so every cluster provides pre-post observations, and switches from control to intervention exposure but not at the same time-point.

This design has been successfully used to implement complex programs and change management involving large-scale programs in many countries. The study also adheres to the various checklists from the EQUATOR network.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 or 65 years of age
* Able to provide informed written consent have been diagnosed with mental health condition, and are ready for discharge.
* Patients should have a mobile device capable of receiving text messages

Exclusion Criteria:

* Patients will be ineligible if they do not meet the above inclusion criteria,
* If they have an addiction disorder but not a mental health diagnosis
* Are not capable of reading text messages from a mobile device or if they know they will be out of town during the 12-month follow-up period.
* Patients are also ineligible if they do not consent to take part in the study,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1132 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in 30 day readmission rate | baseline, 24 weeks, 52 weeks
  Readmission to acute psychiatric care within 30 days of discharge

SECONDARY OUTCOMES:
Change in Clinical Outcomes in Routine Evaluation 10 (CORE-10) scores | baseline, 24 weeks, 52 weeks
  The CORE-10 is a short 10 item easy-to-use assessment measure for common presentations of psychological distress, designed to be used for screening as well as over the course of treatment to track progress. The measure is a shortened version of the 34 item CORE Outcome Measure tool, both of which ask respondents to self-report symptoms over the past week.
Change in EuroQol- 5 Dimension (EQ-5D)scores | baseline, 24 weeks, 52 weeks
  EQ-5D is an instrument which evaluates the generic quality of life
Change in Patient Health Questionnaire (PHQ-9) scores | baseline, 24 weeks, 52 weeks
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression: n The PHQ-9 incorporates the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) depression diagnostic criteria with other leading major depressive symptoms into a brief self-report tool.
Change in Recovery Assessment Scale (RAS)scores | baseline, 24 weeks, 52 weeks
  The RAS is a 20-item measure developed as an outcome measure for program evaluations. Based on a process model of recovery, the RAS attempts to assess aspects of recovery with a special focus on hope and self-determination.
Change in Brief Resilience Scale scores | baseline, 24 weeks, 52 weeks
  The Brief Resilience Scale was created to assess the perceived ability to bounce back or recover from stress. The scale was developed to assess a unitary construct of resilience, including both positively and negatively worded items. The possible score range is from 1 (low resilience) to 5 (high resilience).

OTHER OUTCOMES:
Change in the Reach of the Text4Support | baseline, 24 weeks, 52 weeks
  We will monitor and evaluate changes in the proportion of target population who receive the supportive text messages
Change in the fidelity of the intervention | baseline, 24 weeks, 52 weeks
  We will monitor and evaluate changes in the adherence of peer support workers to the implementation guidelines/protocols
Sustainability of the intervention | 52 weeks
  We will evaluate the proportion of implementation sites who continue implementing the intervention after the active phase of the project
Acceptability of the intervention | 52 weeks
  Using satisfaction surveys, we will evaluate the proportion of participants who found the intervention acceptable

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Agyapong, MD,PhD, Principal Investigator — University of Alberta
Locations (7):
- Canada (7):
  - Royal Alexander Hospital, Edmonton, Alberta
  - Alberta Hospital, Edmonton, Alberta
  - Misericordia Community Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Grey Nuns Hospital, Edmonton, Alberta
  - Northern Lights Regional Health Centre, Fort McMurray, Alberta
  - Foothills Hospital, Calgary

IPD SHARING:
Plan to Share IPD: Yes
Health service utilization information will be collected (for the year prior to admission, and the year post-discharge). This data will include: inpatient admissions and length of stay, readmissions, completed appointments, Emergency Department presentations, Emergency Medical Services use, community services appointments, crisis and urgent service calls, appointment no show rates
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available from the onset of collection till 5 years after the study
Access Criteria: All the hard and electronic copies and other research project related documents will be stored in secure, locked locations and only staff working on this research project will have access to it. Electronic versions of the data will be securely stored in AHS offices.
  The data master list containing identifying data, will be stored separately from other study data, and will only be accessible to the principal investigator and/or their delegate(s)

REFERENCES:
- [Background] Adu MK, Shalaby R, Eboreime E, Sapara A, Nkire N, Chawla R, Chima C, Achor M, Osiogo F, Chue P, Greenshaw AJ, Agyapong VI. Text Messaging Versus Email Messaging to Support Patients With Major Depressive Disorder: Protocol for a Randomized Hybrid Type II Effectiveness-Implementation Trial. JMIR Res Protoc. 2021 Oct 13;10(10):e29495. doi: 10.2196/29495. PMID 34643541
- [Background] Agyapong VIO, Juhas M, Ohinmaa A, Omeje J, Mrklas K, Suen VYM, Dursun SM, Greenshaw AJ. Randomized controlled pilot trial of supportive text messages for patients with depression. BMC Psychiatry. 2017 Aug 2;17(1):286. doi: 10.1186/s12888-017-1448-2. PMID 28768493
- [Background] Shalaby RAH, Agyapong VIO. Peer Support in Mental Health: Literature Review. JMIR Ment Health. 2020 Jun 9;7(6):e15572. doi: 10.2196/15572. PMID 32357127
- [Background] Agyapong VI, Mrklas K, Juhas M, Omeje J, Ohinmaa A, Dursun SM, Greenshaw AJ. Cross-sectional survey evaluating Text4Mood: mobile health program to reduce psychological treatment gap in mental healthcare in Alberta through daily supportive text messages. BMC Psychiatry. 2016 Nov 8;16(1):378. doi: 10.1186/s12888-016-1104-2. PMID 27821096
- [Background] Agyapong VI, Ahern S, McLoughlin DM, Farren CK. Supportive text messaging for depression and comorbid alcohol use disorder: single-blind randomised trial. J Affect Disord. 2012 Dec 10;141(2-3):168-76. doi: 10.1016/j.jad.2012.02.040. Epub 2012 Mar 29. PMID 22464008
- [Derived] Mao W, Shalaby R, Owusu E, Elgendy HE, Agyapong B, Chue P, Silverstone PH, Greenshaw AJ, Li XM, Eboreime E, Vuong W, Ohinmaa A, MacMaster FP, Agyapong V. Predictors of Psychiatric Emergency Department Visits Following Inpatient Discharge: Secondary Analysis of a Stepped-Wedge Cluster Randomized Trial. JMIR Form Res. 2025 Oct 30. doi: 10.2196/79184. Online ahead of print. PMID 41241947
- [Derived] Agyapong VIO, Shalaby R, Agyapong B, Mao W, Owusu E, Elgendy HE, Eboreime E, Silverstone PH, Chue P, Li XM, Vuong W, Ohinmaa A, MacMaster F, Greenshaw AJ. Effectiveness of Text Messages and Text Messages Plus Peer Support on Psychiatric Readmission and Length of Stay: Outcomes From a Quantitative Stepped-Wedge Cluster Randomized Trial. JMIR Ment Health. 2025 Nov 18;12:e81760. doi: 10.2196/81760. PMID 41108215
- [Derived] Owusu E, Mao W, Shalaby R, Elgendy HE, Agyapong B, Eboreime E, Lawal MA, Nkire N, Wei Y, Silverstone PH, Chue P, Li XM, Vuong W, Ohinmaa A, Taylor V, Hilario CT, Greenshaw AJ, Agyapong VIO. The prevalence and correlates of low resilience in patients prior to discharge from acute psychiatric units in Alberta, Canada. BMC Psychiatry. 2025 Mar 27;25(1):295. doi: 10.1186/s12888-025-06704-8. PMID 40148879
- [Derived] Eboreime E, Shalaby R, Mao W, Owusu E, Vuong W, Surood S, Bales K, MacMaster FP, McNeil D, Rittenbach K, Ohinmaa A, Bremault-Phillips S, Hilario C, Greiner R, Knox M, Chafe J, Coulombe J, Xin-Min L, McLean C, Rathwell R, Snaterse M, Spurvey P, Taylor VH, McLean S, Urichuk L, Tzeggai B, McCabe C, Grauwiler D, Jordan S, Brown E, Fors L, Savard T, Grunau M, Kelton F, Stauffer S, Cao B, Chue P, Abba-Aji A, Silverstone P, Nwachukwu I, Greenshaw A, Agyapong VIO. Reducing readmission rates for individuals discharged from acute psychiatric care in Alberta using peer and text message support: Protocol for an innovative supportive program. BMC Health Serv Res. 2022 Mar 12;22(1):332. doi: 10.1186/s12913-022-07510-8. PMID 35279142
- See also: Website documenting evidence from predecessor programs — http://www.resiliencenhope.org/